CLINICAL TRIAL: NCT04590508
Title: A Phase 2 Clinical Trial: Xanthohumol Metabolism and Signature (XMaS) in Crohn's Disease
Acronym: XMaS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Oregon State University (Other); Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Placeholder
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease; IBD; Xanthohumol; Humulus lupulus; Hops
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — xanthohumol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either encapsulated xanthohumol in a rice protein vehicle, or an identical capsule containing vehicle alone.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will occur in up to 8 blocks of 4 based on biological sex. Initial randomization series will be generated using readily available random sequence generators designed to do so. A series of sequential envelopes will be generated, each containing the allocation for one participant. Envelopes will be opaque and signed across the seal. The randomization "code" will be kept in a sealed envelope with a signature across the label and dated the day of creation. Study product and comparator (placebo) will be compounded and placed in identical opaque capsules outside the institution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xanthohumol (Experimental): Participants will take capsules containing 24 mg of xanthohumol in a rice protein vehicle by mouth once daily with the first daily meal.
  Interventions: Drug: Xanthohumol
- Placebo (Placebo Comparator): Participants will receive capsules filled with a rice protein vehicle by mouth once daily with the first daily meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Xanthohumol — The xanthohumol supplement will be administered in a capsule and taken orally.
  Arms: Xanthohumol
Other: Placebo — The placebo will be administered in a capsule and taken orally.
  Arms: Placebo

SUMMARY:
A pilot study to assess the safety and tolerability of an orally administered natural product derived from hops, called xanthohumol, in humans with Crohn's Disease, in order to identify a biological signature of xanthohumol exposure, and to characterize the role of xanthohumol metabolism by intestinal microorganisms in that signature within adults with Crohn's Disease.

DETAILED DESCRIPTION:
This is a double-masked, placebo controlled, randomized clinical trial of xanthohumol, which is a constituent of hops (Humulus lupulus). Hops and its constituents have a long history of use for a variety of conditions. However, knowledge is limited regarding the measurable biological markers of human exposure, and the role of xanthohumol metabolism by microorganisms present in the gut, particularly in individuals with gut pathologies such as Crohn's Disease. This information is necessary for the development of xanthohumol as a potential therapeutic intervention in such conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults 21-50 years of age
* Active Crohn's disease not in remission based on a CDAI score >150
* Willing to take isolated Xanthohumol as a dietary supplement for 8 weeks
* Willing to have blood drawn bi-weekly and fast for 10-12 hours before blood draws
* Willing and able to collect bi-weekly stool samples at home
* Willing and able to collect a 24-hour urine sample before each study visit
* Able to speak, read and understand English
* Must be able to provide written informed consent
* Non-smokers (including tobacco and Cannabis products, combusted or vaporized)
* For individuals of child-bearing potential, willingness to use an intrauterine device (IUD) or two other concurrent forms of birth control (e.g., 2 of the following categories: condoms, spermicide-containing gels, films or sponges; and/or vaginal rings) to prevent pregnancy while enrolled

Exclusion Criteria:

* Highly variable dosing of anti-inflammatory medications (dose changes more than 1x per week)
* Currently or recent (within last 14 days) taking any dietary supplements containing xanthohumol, flavonoids, or other known "anti-inflammatories" including: curcumin, turmeric, fenugreek, hops, rosemary, ginger, white willow, devil's claw, fish oil (doses>1 g/day), or quercetin. Candidates will be given the option to "wash out" for 14 days and re-contact the study team.
* Consumption of more than 1 beer per day.
* Currently receiving intravenous nutrition support therapy (or within the last 14 days)
* Currently taking anti-coagulant or anti-platelet prescription medications (or they were taken within the last 14 days)
* Currently taking antibiotic, antiparasitic, or antifungal medications orally or intravenously (or they were taken within the last 14 days)
* Initiation of or changes to supplements or medications within 14 days prior to screening.
* Initiation of or changes to an exercise regimen within 14 days prior to screening.
* Initiation of or changes to a food plan within 14 days prior to screening.
* Current involvement or within 14 days prior to screening of a significant diet or weight loss program (such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs) or very low-calorie liquid diet programs (such as Optifast, Medifast, and/or HMR)
* Hospitalization (for any reason other than a scheduled medical procedure) within 3 months prior to screening
* Gastrointestinal surgery within 3 months prior to screening
* Malignancy within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
* Women who are lactating, pregnant or planning pregnancy within the next four months
* Typical intake of more than 2 alcohol-containing beverages per day, more than 14 per week, or more than 4 in any single day within the past 14 days.
* Smoking tobacco or nicotine products (combusted or vaporized)
* Use of illicit drugs/substances (such as but not limited to cocaine, phencyclidine (PCP), and methamphetamine) within 14 days of screening
* Use of inhaled or ingested Cannabis products, including Cannabidiol (CBD)
* Currently participating in another interventional research study, or participated in another interventional research study within 14 days of screening
* Do not have an active primary care provider or specialist (i.e., gastroenterologist) managing their CD

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline: Aspartate aminotransferase (AST) | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Aspartate aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as: % abnormal, % new abnormals, and mean change from baseline.
Change from Baseline:Alanine aminotransferase (ALT) | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Alanine aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as: % abnormal, % new abnormals, and mean change from baseline.
Change from Baseline: gamma-Glutamyl transferase (GGT) | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Gamma-glutamyl transferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as: % abnormal, % new abnormals, and mean change from baseline.
Change from Baseline: Estimated glomerular filtration rate | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Glomerular filtration rate is estimated based on blood creatinine concentration per standard nephrology practice. Reported as: % abnormal, % new abnormals, and mean change from baseline.
Change from Baseline: Blood urea nitrogen to creatinine ratio | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Blood urea nitrogen:creatinine is a ratio of serum concentrations of two compounds associated with renal function. Reported as: % abnormal, % new abnormals, and mean change from baseline.
Change from Baseline: Complete blood count | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Enumeration of the various subtypes of blood cells (i.e., red blood cells, white blood cells, and platelets), plus indices including mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), and hemocrit. Reported as: % abnormal, % new abnormals, and mean change from baseline.

SECONDARY OUTCOMES:
Change from Baseline: Composite Symptoms: Crohn's Disease Activity Index (CDAI) | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  The Crohn's Disease Activity Index or CDAI is frequently used to assess disease severity. It gives a score ranging from 0 to over 600, based on a diary of symptoms kept by the patient for 7 days, and other measurements such as the patient's weight and haematocrit. A CDAI score of less than 150 is considered to be remission, a score greater than 220 is considered to define moderate to severe disease, and a score greater than 300 is considered to be severe disease. Most major research studies on medications in Crohn's disease define response as a fall of the CDAI of greater than 70 points.
Change from Baseline: Change in fecal calprotectin levels | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Fecal calprotectin, a protein associated with gut inflammation and irritable gut syndrome, will be measured by enzyme-linked immunosorbent assay, and expressed as mean change over time from baseline.
Change from Baseline: Change in plasma inflammatory markers (pg/mL) | 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Circulating pro-inflammatory cytokine concentrations (tumor necrosis factor (TNF)-α, interleukin (IL)-1β, IL-2, IL-6, IL-8, IL-10, , and IL-12p70), will be measured simultaneously with a flow cytometry-based multiplex assay. The results will be expressed as change from baseline over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND/MPH, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use the University of California San Diego (UCSD) Metabolomics Workbench for sharing metabolomics datasets and results (including raw data matrices, platform information, and associated metadata).
  For activity-based proteomics data, we will use PRIDE or the MassIVE data repository at UCSD.
  Nucleic acid sequence data will be submitted to the National Center for Biotechnology Information (NCBI) Short Read Archive.
  Gene expression data will be submitted to Gene expression Omnibus at NCBI. Microbiome metadata will be deposited into database of Genotypes and Phenotypes.
  Metagenomic nucleic acid sequence data will additionally be deposited in Metagenomic Rapid Annotations using Subsystems Technology (MG-RAST) at Argonne National Laboratory, along with associated metadata.
  Microbiome summary files (e.g., tables cataloging: sample metadata, taxon or protein family abundances across samples) publicly available through github.
Supporting Information: Study Protocol
Time Frame: We will share our data no later than on acceptance of the first publication of the findings from the respective data set(s).

REFERENCES:
- [Derived] Langley BO, Ryan JJ, Phipps J, Buttolph L, Bray B, Aslan JE, Metz TO, Stevens JF, Bradley R. Xanthohumol microbiome and signature in adults with Crohn's disease (the XMaS trial): a protocol for a phase II triple-masked, placebo-controlled clinical trial. Trials. 2022 Oct 22;23(1):885. doi: 10.1186/s13063-022-06782-z. PMID 36273173